CLINICAL TRIAL: NCT00346385
Title: A Phase I, Open-Label, Dose Escalation Study of Daily Dosing With BB-10901
Brief Title: BB-10901 in Treating Patients With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000491231; IMMUNO-C10/IVB/002; IMGN-002; MDA-2004-0557; NCT00625287 (obsolete NCT alias)
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Ovarian Cancer; Merkel Cell Carcinoma; SCLC
Keywords: recurrent small cell lung cancer; merkel cell carcinoma; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Merkel Cell; Small Cell Lung Carcinoma | interventions — lorvotuzumab mertansine

INTERVENTIONS:
Drug: BB-10901 — dose escalation study, dose will vary per cohort. patients will receive an IV infusion once every three weeks.
  Other Names: IMGN901

SUMMARY:
RATIONALE: Monoclonal antibodies, such as BB-10901, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase I trial is studying the side effects and best dose of BB-10901 in treating patients with relapsed or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of BB-10901
* Determine the maximum tolerated dose of this drug in these patients.

Secondary

* Determine the pharmacokinetics of this drug in these patients.
* Determine the efficacy of this drug in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study.

Patients receive BB-10901 IV over 40 minutes once daily on days 1-3.* Treatment repeats every 21 days

NOTE: *Patients who do not tolerate 3 consecutive daily infusions of BB-10901 may receive infusions of BB-10901 on 3 alternate days, upon approval by the investigator and/or the independent Safety Review Board.

Cohorts of 4-6 patients receive escalating doses of BB-10901 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 4-6 patients experience dose-limiting toxicity in course 1. Up to 40 patients are treated at the MTD.

After completion of study treatment, patients are followed for short term and long term follow up and survival.

PROJECTED ACCRUAL: Approximately 100 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS During Dose Escalation:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Small cell lung cancer (SCLC)
  * Other pulmonary tumors of neuroendocrine origin, including neuroendocrine carcinoma or non-SCLC with neuroendocrine features
  * Non-pulmonary small cell carcinoma
  * Metastatic carcinoid tumor
  * Other CD56-positive solid tumor
* Diagnoses other than SCLC must have confirmation of tumor CD56 expression before study entry
* Relapsed or refractory disease
* Must have received at least 1 but no more than 3 prior chemotherapy regimens* and recovered from any acute toxicities

  * No prior chemotherapy for carcinoid or neuroendocrine tumors

DISEASE CHARACTERISTICS During MTD Expansion:

* Relapsed or refractory Small cell lung cancer (SCLC)
* Metastatic Merkel Cell carcinomas
* Ovarian carcinomas

At the MTD:

SCLC patients must have received one, but no more than 1 prior chemotherapy regimen Merkel and Ovarian patients must have received at least one prior chemotherapy regimen. Ovarian patients must have received at least one platinum-based regimen.

* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* No uncontrolled carcinoid syndrome (e.g., flushing, uncontrolled diarrhea, labile blood pressure)
* No active brain metastases; no evidence of active disease and no requirement for anticonvulsant medications or steroids.

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 months
* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Bilirubin ≤ 3 times ULN
* No rapidly rising liver function tests (LFTs)
* Pancreatic function, amylase and lipase within upper limit of normal.
* No significant residual neurological or cardiac toxicity ≥ grade 2 after prior chemotherapy
* No myocardial infarction within the past 6 months
* No unstable angina pectoris
* No uncontrolled congestive heart failure
* No uncontrolled arrhythmia
* No severe aortic stenosis
* No history of multiple sclerosis or other demyelinating disease
* No Eaton-Lambert syndrome (para-neoplastic syndrome)
* No history of hemorrhagic stroke
* No CNS injury with residual neurologic deficit
* No ischemic stroke within the past 6 months
* No history of pancreatitis
* No current active infection or history of recurrent infection with varicella-zoster virus (shingles) or cytomegalovirus
* No other concurrent serious infection
* No chronic alcoholism
* No other concurrent illness or condition that would interfere with study outcome
* No other malignancy within the past 3 years except adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No known recent biochemical or clinical evidence of pancreatitis or extensive metastatic disease involving the pancreas

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Total cumulative dosage of prior anthracycline treatment must not exceed threshold for cardiotoxicity
* No known hypersensitivity to previous monoclonal antibody therapy
* More than 4 weeks since prior and no concurrent chemotherapy or radiotherapy
* More than 4 weeks since prior and no other concurrent investigational agents
* At least 4 weeks since prior and no concurrent surgery
* No other concurrent antineoplastic treatment, including immunotherapy or steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2002-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by toxicity evaluation and prothrombin time assessments | these tests will be conducted at various timepoints during a patients participation in the trial

SECONDARY OUTCOMES:
Pharmacokinetics assessed by measuring intact conjugate and total huN901 antibody concentration for each time point and dose level | PK is assessed during the first cycle (21 days) of a patients participation
Efficacy assessed by measuring response (complete or partial response) and biomarker levels of neuron-specific enolase and soluble neural cell adhesion molecules (NCAM) | efficacy is assessed every 2 cycles during a patients participation while other blood tests are taken during every cycle

CONTACTS AND LOCATIONS:
Overall Officials: Paul C. Lorigan, MD, Study Chair — The Christie NHS Foundation Trust
Locations (9):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - Nevada Cancer Institute, Las Vegas, Nevada
  - The Ohio State University Cancer Center and Research Institute, Columbus, Ohio
  - Oklahoma University, Oklahoma City, Oklahoma
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- United Kingdom (3):
  - Christie Hospital NHS Trust, Manchester, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England